CLINICAL TRIAL: NCT00247325
Title: Renal Toxicity Evaluation and Comparison Between Visipaque (Iodixanol) and Hexabrix (Ioxaglate) in Renal Insufficiency Undergoing Coronary Angiography: The RECOVER Study, A Randomized Controlled Trial
Brief Title: RECOVER:Comparison of Renal Toxicity Between Visipaque(Iodixanol)and Hexabrix(Ioxaglate)in Renal Insufficiency Undergoing Coronary Angiography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 144-가-24; 144-가-24
Record Dates: First submitted 2005-10-31; First posted 2005-11-01 (Estimated); Last update posted 2006-11-30 (Estimated); Status verified 2005-01

CONDITIONS: Kidney Failure
Keywords: Kidney failure; Contrast media; Iodixanol; Ioxaglate
MeSH Terms: conditions — Renal Insufficiency

INTERVENTIONS:
Drug: Iodixanol(Drug)

SUMMARY:
In the treatment of coronary heart disease which is the major cause of heart attack, direct mechanical treatment with catheters such as the coronary angiography,coronary balloon intervention and stenting intervention are the mainstay of therapy in recent years. In that procedures, we should use the contrast media, and it may cause kidney toxicity especially in the patients with underlying kidney disease and decreased kidney function. We intended to find out which contrast agent has less kidney toxicity in the catheter based treatment of coronary arterial diseases in patients with underlying decreased kidney function

DETAILED DESCRIPTION:
Iodixanol, a nonionic, dimeric, iso-osmolar contrast medium (IOCM), may be less nephrotoxic than nonionic, monomeric, low-osmolar contrast media (LOCMs) in high-risk patients. We compared the nephrotoxicity of iodixanol with that of ioxaglate, an ionic, dimeric LOCM, in patients with renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* creatinine clearance rates ≤60 mL/min using the Cockcroft-Gault formula
* Patients who undergo coronary catheterization
* Age of 19 or over 19.

Exclusion Criteria:

* pregnancy
* lactation
* having received contrast media within 7 days of study entry
* emergent coronary angiography
* acute renal failure
* end-stage renal disease requiring dialysis
* history of hypersensitivity reaction to contrast media
* cardiogenic shock
* pulmonary edema
* multiple myeloma
* mechanical ventilation
* parenteral use of diuretics
* use of N-acetylcysteine
* use of metformin or nonsteroidal anti-inflammatory drugs within 48 hours of the procedure.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-01; Study Completion 2004-12

PRIMARY OUTCOMES:
Incidence of contrast induced nephropathy, defined as either a relative increase in serum creatinine from baseline of >=25% or an absolute increase of >=0.5mg/dL(44.2µmol/L) during days 1 and 2

SECONDARY OUTCOMES:
proportion of patients exhibiting an increase in serum creatinine of >=0.5mg/dL(44.2µmol/L), the proportion with a >=1.0 mg/dL(88.4µmol/L) increase in serum creatinine, and the mean peak increase in serum creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Soo Kim, M.D., Ph.D., Study Director — Seoul National University Hospital, Cardiovascular Center; Byung-Hee Oh, M.D., Ph.D., Study Chair — Seoul National University Hospital, Internal Medicine/ Cardiovascular Center; Sang-Ho Jo, M.D., Principal Investigator — Seoul National University Hospital, Cardiovascular Center
Locations (1):
- Seoul National University Hospital , Cardiovascular Center, Seoul, South Korea

REFERENCES:
- [Result] Jo SH, Youn TJ, Koo BK, Park JS, Kang HJ, Cho YS, Chung WY, Joo GW, Chae IH, Choi DJ, Oh BH, Lee MM, Park YB, Kim HS. Renal toxicity evaluation and comparison between visipaque (iodixanol) and hexabrix (ioxaglate) in patients with renal insufficiency undergoing coronary angiography: the RECOVER study: a randomized controlled trial. J Am Coll Cardiol. 2006 Sep 5;48(5):924-30. doi: 10.1016/j.jacc.2006.06.047. Epub 2006 Aug 17. PMID 16949481